CLINICAL TRIAL: NCT03802942
Title: Prevention of Hypoglycemia Among Diabetes Patients Admitted to Internal Medicine Departments, by Means of a Designated Nutritional Care Program
Brief Title: Prevention of Hypoglycemia Among Diabetes Patients Admitted to Internal Medicine Departments With Nutritional Care
Acronym: MENU-DM
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eyal Leibovitz (Other)
Collaborators: Abbott Nutrition (Industry)
Responsible Party: Sponsor-Investigator, Eyal Leibovitz, Chair, Internal medicine unit B, Laniado hospital, Yoseftal Hospital
Organization: Yoseftal Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EL001MENU-DM
Record Dates: First submitted 2019-01-08; First posted 2019-01-14 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Hypoglycemia; Malnutrition; Diabetes
Keywords: hypoglycemia; diabetes mellitus; malnutrition
MeSH Terms: conditions — Hypoglycemia; Malnutrition; Diabetes Mellitus | interventions — Glucerna

STUDY DESIGN:
Intervention Model Description: Randomized open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glucerna (Experimental): 2 bottles of Glucerna per day (237 ml per bottle for a total of 474 ml/d) on top of the meal plan supplied by the hospital.
  Interventions: Dietary Supplement: Glucerna
- Control (No Intervention): Regular meal plan supplied by the hospital

INTERVENTIONS:
Dietary Supplement: Glucerna — 1 bottle in the morning with breakfast and 1 bottle in the evening with dinner
  Arms: Glucerna

SUMMARY:
This is a prospective randomized study to evaluate the efficacy of nutritional intervention for the prevention of hypoglycemia among diabetes patients with low albumin level that are admitted to internal medicine units, regardless of the reason for admission. All patients suitable for participation in the study will be asked to participate and be randomized to the interventional arm or the control arm.

After admission to the internal medicine unit, eligible patients will be asked to participate in the study. After signing an informed consent form, patients will be randomized to the treatment or control arms. For patients allocated to the treatment arm, the physician in charge will prescribe 2 portions of GlucernaTM per day as part of the treatment protocol. The nurse in charge of the patient (at either the morning or evening shifts) will make sure the patient is receiving and consuming the ONS.

For every patient included in the interventional arm, 2 bottles of GlucernaTM will be supplied to the patient, one at 08:00 with the morning medications, and one at 16:00 with the evening medications. For clarification purposes, the GlucernaTM will be supplied on top of the designated meal plan, as "over-feeding". Evaluation of adequate ONS consumption will be performed 2-3 hours after the dispensing of the ONS (at 10:00-11:00 and 19:00-21:00), and the amount consumed will be documented.

Patients in the control arm will receive no oral nutritional supplementation, and their caloric intake will be composed of the food supplied by the hospital. Other analysis will be considered usual care. Additional diet consultations as requested by the medical staff will constitute usual care, and the patient will continue the study.

The duration of ONS treatment will be the entire length of hospital stay. Upon discharge, a recommendation to continue nutritional care will be added to the patients' discharge letters but no oral nutritional supplement (ONS) will be prescribed or dispensed.

Following discharge, a 30-day follow-up call will be made to ascertain whether the patient is alive, whether the patient was re-admitted or re-hospitalized, and the usage of ONS prescribed by the family/general practitioner that was consumed after the hospital discharge.

DETAILED DESCRIPTION:
1.2 Definitions: A. Hypoglycemia: a blood glucose level of 70 mg/dL or lower, regardless of symptoms B. Hypoalbuminemia: Albumin level below 3.5 g/dL upon admission to the hospital C. Adequate nutritional consumption: the consumption of at least half of the oral nutritional supplements D. Target population: Diabetes patients admitted to internal medicine units that have baseline hypoalbuminemia upon admission.

This is a prospective randomized study to evaluate the efficacy of nutritional intervention for the prevention of hypoglycemia among diabetes patients with low albumin level that are admitted to internal medicine units, regardless of the reason for admission. All patients suitable for participation in the study will be asked to participate and be randomized to the interventional arm or the control arm.

After admission to the internal medicine unit, eligible patients will be asked to participate in the study. After signing an informed consent form, patients will be randomized to the treatment or control arms. For patients allocated to the treatment arm, the physician in charge will prescribe 2 portions of GlucernaTM per day as part of the treatment protocol. The nurse in charge of the patient (at either the morning or evening shifts) will make sure the patient is receiving and consuming the ONS.

2.3 Study population: All adult patients admitted to internal medicine units of the Wolfson Medical Center that will participate in the study. The admission to the unit can be either from the ER or as a transfer from other departments in the hospital.

Inclusion and Exclusion criteria specified above.

Drop-out criteria A. Patients in need of mechanical nutritional support (same as above), as a complication of the hospitalization.

B. Patients that have a designated nutritional care program recommended by the unit's dietician that includes ONS. For clarification purposes, fortification of the meal plan by changing the food items (i.e. low sugar items, high fat/protein and or etc.) will not be considered a drop-out indication, as long as ONS are not part of the intervention.

C. Patients with undocumented albumin level for the first 72 hours of the hospitalization to the internal medicine unit.

D. Patients that were enrolled in the study but were transferred from the internal medicine department to a different unit of treatment during the hospitalization. For clarification purposes, transfer to interventional radiology, interventional cardiology or any other units for a specific procedure is not considered a dropout criteria, as long as the patient is back in the internal medicine unit within 24-48 hours of the procedure.

2.4 Interventional program Interventional arm A. For every patient included in the interventional arm, 2 bottles of GlucernaTM will be supplied to the patient, one at 08:00 with the morning medications, and one at 16:00 with the evening medications. For clarification purposes, the GlucernaTM will be supplied on top of the designated meal plan, as "over-feeding".

B. Evaluation of adequate ONS consumption will be performed 2-3 hours after the dispensing of the ONS (at 10:00-11:00 and 19:00-21:00), and the amount consumed will be documented.

C. Patients in the intervention arm that will be unwilling to consume the ONS will not drop out of the study, but rather the follow-up will continue as usual (ITT design). The ONS will be offered every day, twice a day, regardless of the answer and the amount consumed. For patients that decline, the reason for lack of consumption will be documented.

D. The duration of ONS treatment will be the entire length of hospital stay. Upon discharge, a recommendation to continue nutritional care will be added to the patients' discharge letters but no ONS will be prescribed or dispensed.

Control arm A. Patients in the control arm will receive no oral nutritional supplementation, and their caloric intake will be composed of the food supplied by the hospital. Other analysis (i.e. malnutrition screen, blood tests etc.) will be considered usual care. Additional diet consultations as requested by the medical staff will constitute usual care, and the patient will continue the study, as long as no additional ONS are prescribed as part of the treatment plan (criteria 2 of the drop-out criteria).

B. Upon discharge, a recommendation to continue nutritional care will be added to the patients' discharge letters but no ONS will be prescribed or dispensed.

Post discharge, all patients

Following discharge, a 30-day follow-up call will be made to ascertain key points:

A. Whether the patient is alive B. Whether the patient was re-admitted or re-hospitalized C. Usage of ONS prescribed by the family/general practitioner that was consumed after the hospital discharge.

3.1 informed consent The study will seek the approval of the local Institutional Review Board (IRB) as an interventional study. All patients participating (either in the treatment or control arms) will sign an informed consent upon study inclusion.

3.2 Data recording For each patient, a paper case report form (CRF) will be produced. The patient data recorded in the CRFs will include the following information A. demorgaphic data A.1. Age, sex, marital status B. Reason for admission, one or more of the following (multiple selection) B.1. Infection (pneumonia/other) B.2. Acute coronary disease B.3. Acute cerebrovascular accident (CVA) (all types) C Patient co-morbidities - one or more of the following (multiple selection) C.1. Hypertension C.2. Hyperlipidemia C.3. Chronic renal failure C.4. Cerebrovascular disease C.5. Coronary artery disease C.6. Congestive heart failure C.7. Chronic obstructive pulmonary disease C.8. Dementia (all stages) D Nutritional assessment - all the following (mandatory for all patients) D.1. Subjective global assessment D.2. Height (or knee height for patients that cannot be measured) D.3. Weight (or mid arm circumference for patients that cannot be measured) E Admission laboratory values - all the following (mandatory for all patients) E.1. Hemoglobin level E.2. White blood cell count E.3. C-Reactive protein E.4. Albumin and pre-albumin E.5. HbA1c E.6. Creatinine E.7. Recording of all glucose measurements F Medication plan (mandatory for all patients) F.1. Lipid lowering drugs (any type any dose) - y/n F.2. Antibiotic treatment (any type any dose) - y/n: for clarification: any type of antibiotic treatment given orally or by injection (IM, IV, intra-articular etc.). Topical antibiotics (either ointment or solution) will not be recorded.

F.3. Gluco-corticoid treatment (any type any dose) - y/n: for clarification: any type of gluco-corticoid treatment given orally or by injection (IM, IV, intra-articular etc.). Topical steroid treatment (either ointment or solution) will not be recorded.

F.4. Glucose lowering medications F.4.1. Insulin treatment (any type any dose) - y/n F.4.2. Glucagon-like peptide-1/Dipeptidyl peptidase-4 inhibitors (GLP1/DPP4i) (any type any dose) - y/n F.4.3. Metformin (any type any dose) - y/n F.4.4. Other (any type any dose) - y/n G.1. Meal consumption according to nutrition day analysis - daily 3 meals per day G.2. Glucerna ONS consumption - 2 bottles dispensed. Each day an estimation of each H Prognostic criteria H.1. Length of hospital stay - post discharge H.2. In-hospital and/or 30 day mortality (if applicable) H.3. 30-day readmission (if applicable).

Follow-up call For prognostic criteria assessment, a phone call will be made 30 days after discharge to ascertain survival and need for hospitalization. Readmission will be any and all referrals to an emergency room. A distinction will be made if the referral to the ER was followed by an admission to the hospital. The reason for readmission or re-hospitalization will not be recorded. For clarification purposes an admission for an elective surgery or procedure (i.e. coronary angiogram), or an elective admission for continuing care will not be considered a readmission.

ELIGIBILITY:
Inclusion Criteria:

* admission to internal medicine units &
* Diabetes mellitus type 2 &
* Admission serum-albumin level below 3.5 gr/dL.

Exclusion Criteria:

* nasogastric [NG] tube
* percutaneous endoscopic gastrostomy [PEG]
* feeding jejunostomy
* total parenteral nutrition [TPN]
* chemotherapy or immunotherapy for malignancy during the past 6 months
* Malignancy with life expectancy of less than 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Total number of patients with at least 1 documented low (equal or below 70 mg/dL) glucose levels | During the entire hospital stay, estimated up to 60 days
  The number of patients with at least 1 documented glucose levels equal or below 70 mg/dL for the entire study arm

SECONDARY OUTCOMES:
Total number of documented low (equal or below 70 mg/dL) glucose levels | During the entire hospital stay, estimated up to 60 days
  The number of documented glucose levels equal or below 70 mg/dL for the entire study arm
Length of hospital stay | During the entire hospital stay, estimated up to 60 days
  Average length of hospital stay in days of the patients according to study arm
In-hospital and 30-day mortality rates | Estimated up to 90 days
  Death of patients occuring during hospitalization or within 30 days from discharge of patients according to study arm
30-day readmission rate | During the first 30 days from discharge
  Referral to the Emergency room or readmission to the hospital within 30 days from discharge

CONTACTS AND LOCATIONS:
Overall Officials: Eyal Leibovitz, MD, Principal Investigator — Yoseftal Hospital
Locations (2):
- Israel (2):
  - Yoseftal hospital, Eilat
  - Wolfson Medical Center, Holon

IPD SHARING:
Plan to Share IPD: No